CLINICAL TRIAL: NCT07140055
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Single-ascending Dose and Multiple-ascending Dose (SAD and MAD) Trial to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Novel Glucagon-like Peptide-1 Receptor Agonist (GLP-1RA) BLX-7006 in Healthy Adults With a Body Mass Index (BMI) of 20 - 35 kg/m2
Brief Title: A Research Study to Evaluate BLX-7006 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biolexis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BLX-7006-CLN-001
Record Dates: First submitted 2025-08-04; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Normal Healthy Volunteer; Safety After Oral Intake
Keywords: Obesity; Type 2 Diabetes; Metabolic Disorders; Normal Healthy Volunteer
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLX-7006 Oral Dose (Experimental): Participants will receive oral BLX-7006 as a single dose (in Part 1 or 2) or once daily for 7 days (in Part 3).
  Interventions: Drug: BLX-7006
- Placebo to match BLX-7006 (Placebo Comparator): Participants will receive an oral placebo that looks like BLX-7006 but does not contain active drug as a single dose (in Part 1 or 2) or once daily for 7 days (in Part 3).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLX-7006 — BLX-7006 Single or Multiple doses administered orally as a tablet
  Arms: BLX-7006 Oral Dose
Drug: Placebo — Participants will receive matching placebo of BLX-7006 for each of the oral cohorts.
  Arms: Placebo to match BLX-7006

SUMMARY:
This study will test an oral medicine called BLX-7006, which acts like the hormone Glucagon-like Peptide-1 (GLP-1) to help control blood sugar and body weight. Current GLP-1 medicines are given by injection. This study will see if BLX-7006 is safe, how the body processes it, and whether food changes how it is absorbed. The main goal is to see if BLX-7006 is safe and well tolerated. Secondary objectives of the study will measure how BLX-7006 moves through the body after an oral dose, including how quickly it is absorbed, how long it stays in the blood, and how the body removes it. It will also look at how the drug affects the body by looking at markers of glucose metabolism.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and the effect of food on the PK of BLX-7006, a novel oral small-molecule GLP-1 receptor agonist, in healthy adult volunteers. The study consists of three parts: single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) assessments.

Study Rationale and Objectives:

BLX-7006 is being developed as an oral alternative to currently available injectable GLP-1 receptor agonists used for the treatment of metabolic diseases such as type 2 diabetes mellitus and obesity. Oral delivery of BLX-7006 may improve convenience and treatment adherence while maintaining the metabolic benefits of GLP-1 agonism. This Phase 1 study is designed to characterize the initial safety profile, define the PK properties of BLX-7006, evaluate preliminary PD biomarkers of glucose metabolism, and determine the impact of a high-fat meal on drug absorption.

Study Design Overview:

The study will enroll approximately 76 healthy adults across three sequential parts.

Part 1: Single Ascending Dose (SAD) This is a randomized, double-blind, placebo-controlled, sequential SAD study in up to four cohorts (approximately 8 participants per cohort; 6 active, 2 placebo). Doses will escalate sequentially following review of blinded safety, tolerability, PK, and PD data by a Safety Review Committee (SRC). A sentinel dosing approach will be used for each cohort (1 active, 1 placebo) prior to dosing the remainder of the cohort. Participants will be confined in the clinical research unit (CRU) for approximately 4 days for safety monitoring, PK and PD blood sampling, and will return for an end-of-study (EOS) visit on Day 8. SAD data will inform dose selection for the FE and MAD parts of the study.

Part 2: Food Effect (FE) This is an open-label, randomized, 2-period, 2-sequence crossover study designed to evaluate the effect of a high-fat, high-calorie meal on the PK of a single oral dose of BLX-7006. A single cohort of 12 participants will receive BLX-7006 under both fasted and fed conditions, with a 7-day washout between doses. Participants will be confined for approximately 4 days in each period, with safety, PK, and PD assessments performed throughout. The SRC may adjust the washout interval or timing of assessments based on PK results from the SAD cohorts to ensure adequate elimination between periods.

Part 3: Multiple Ascending Dose (MAD) This is a randomized, double-blind, placebo-controlled, sequential MAD study in up to four cohorts (approximately 8 participants per cohort; 6 active, 2 placebo). Participants will receive BLX-7006 or placebo orally once daily for 7 days. Participants will be confined from Day -1 through approximately Day 10 for dosing, safety assessments, and PK/PD sampling, with an EOS visit on Day 14. Dose escalation to subsequent MAD cohorts will occur following review of blinded safety, PK, and PD data by the SRC.

Safety Monitoring:

Safety will be evaluated throughout the study by monitoring adverse events (AEs), clinical laboratory tests, vital signs, 12-lead electrocardiograms (ECGs), and physical examinations. Sentinel dosing and SRC reviews between cohorts are incorporated to minimize risk.

Pharmacokinetic and Pharmacodynamic Assessments:

Blood samples will be collected to characterize single- and multiple-dose PK parameters of BLX-7006, including maximum concentration (Cmax), time to maximum concentration (Tmax), area under the curve (AUC), half-life (t½), and apparent clearance. PD endpoints will include biomarkers of glucose metabolism and insulin production. The FE part will compare PK parameters between fasted and fed states.

Dose Escalation and Cohort Progression:

The SRC will review cumulative safety, tolerability, PK, and PD data after each cohort before escalating to the next dose level. The number of cohorts may be reduced based on emerging data. The FE and MAD parts may proceed in parallel with later SAD cohorts once predefined safety criteria are met.

The results of this study will provide the initial clinical safety and PK/PD profile of BLX-7006, including preliminary assessment of food effect, to support future clinical development in populations with metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 18-65 years, BMI 20-35 kilograms/meter² (kg/m²), weight ≥50 kilograms (kg).
* Normal or clinically acceptable labs, vital signs
* HbA1c <6.5%, non-fasting glucose 4.0-7.8 milimol/Liter (mmol/L)
* Willing to follow contraception requirements, avoid alcohol, nicotine, and blood donation per protocol, and comply with all study visits and procedures.

Exclusion Criteria:

* History of diabetes, clinically significant cardiovascular, hepatic, renal, gastrointestinal, psychiatric, or neurologic disease, or abnormal labs/Echocardiograms (ECG) deemed clinically relevant.
* Prior gastrointestinal (GI) surgery affecting absorption (e.g., gastric bypass) or chronic GI disorders.
* History or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia type 2 (MEN2); malignancy within 5 years (except treated basal cell or in situ cervical cancer).
* History of severe allergic reactions, seizures, or psychiatric hospitalization; positive drug, alcohol, or cotinine test.
* Use of prescription drugs, Over the counter (OTC) /herbal supplements
* Participation in another clinical trial or blood donation within 30 days (or 5 half-lives of prior drug).
* Any condition or history that may compromise safety, study conduct, or compliance, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced Adverse Events (AEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-7006 administration will be evaluated based on the incidence of adverse effects in subjects, as assessed according to CTCAE v5.0. The number of participants who experience an AE will be reported.
Number of participants who experienced Serious Adverse Events (SAEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-7006 administration will be evaluated based on the incidence of SAE in subjects, as assessed according to CTCAE v5.0. The number of participants who experience a SAE will be reported.
Number of participants who experienced Treatment-Related Adverse Avents (TRAEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-7006 administration will be evaluated based on the incidence of TRAEs in subjects, as assessed according to CTCAE v5.0. The number of participants who experience a TRAE will be reported.

SECONDARY OUTCOMES:
Assess maximum observed drug concentration (Cmax) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-7006 in single, food effect, and multiple ascending doses in healthy adults
Assess time to maximum concentration (Tmax) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-7006 in single, food effect, and multiple ascending doses in healthy adults
Assess the area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-7006 in single, food effect, and multiple ascending doses in healthy adults
Assess the area under the concentration curve from time 0 to the last quantifiable concentration (AUClast) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-7006 in single, food effect, and multiple ascending doses in healthy adults
Assess half-life (t½) plasma concentration | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-7006 in single, food effect, and multiple ascending doses in healthy adults
Serum fructosamine levels | Up to 14 days after last dose in each cohort
  Evaluate the effect of single and multiple oral doses of BLX-7006 on serum fructosamine levels
Insulin levels | Up to 14 days after last dose in each cohort
  Evaluate the effect of single and multiple oral doses of BLX-7006 on insulin levels
C-peptide levels | Up to 14 days after last dose in each cohort
  Evaluate the effect of single and multiple oral doses of BLX-7006 on C-peptide levels
Glucagon levels | Up to 14 days after last dose in each cohort]
  Evaluate the effect of single and multiple oral doses of BLX-7006 on glucagon levels

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane Clinic, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No